CLINICAL TRIAL: NCT04714736
Title: Renal Insufficiency Following Contrast Media Administration Trial IV: Contrast Media Volume Control for Limiting Contrast-Induced Acute Kidney in Acute Coronary Syndrome.
Brief Title: DyeVert System and Contrast-induced Acute Kidney Injury
Acronym: REMEDIALIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Mediterranea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NCT006
Record Dates: First submitted 2021-01-10; First posted 2021-01-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Contrast-induced Acute Kidney Injury; Acute Coronary Syndromes
Keywords: acute kidney injury; Device: DyeVert™ system; percutaneous coronary intervention
MeSH Terms: conditions — Acute Coronary Syndrome; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Patients included into the study will be treated according to the following strategy. Patients will receive intravenous 0.9% sodium chloride as soon as in the catheterization laboratory. The hydration regimen will be defined according to the hemodynamic conditions, as defined below. The patients will be then randomized into two groups: 1) DyeVert group, and 2) Control group.
Who Masked: Participant
Masking Description: Patients will be then randomized into 2 groups: 1) DyeVert group, and 2) Control group.
  DyeVert group: injection will be handled by the DyeVert system. Control group: injection will be carried out by manual injection syringe. Patients don't know the arm in which they are assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DyeVert group (Active Comparator): Patients will receive intravenous 0.9% sodium chloride as soon as in the catheterization laboratory. The hydration regimen will be defined according to the hemodynamic conditions and modulated according to the left ventricular end diastolic pressure (LVEDP). During the PCI the CM injection will be handled by the DyeVert TM system.
  Interventions: Device: Coronary angiography using DyeVert system
- Control group (Sham Comparator): Patients will receive intravenous 0.9% sodium chloride as soon as in the catheterization laboratory. The hydration regimen will be defined according to the hemodynamic conditions and modulated according to the left ventricular end diastolic pressure (LVEDP). During the PCI the CM injection will be carried out by a conventional manual injection syringe. Strategies for limiting CM volume are:
  1. angiograms will be performed with injection of contrast using a 3-cm 3 syringe; this provides strict control of CM delivery by limiting the volume of contrast that can be administered in a single injection;
  2. catheters with sideholes will be strictly avoided during percutaneous intervention;
  3. when exchanging catheters, unused contrast is withdrawn from the catheter lumen (e.g., by back-bleeding through an opened ''Y''-connector or by aspirating residual contrast from the catheter using a syringe)
  4. ''tests'' with ''puffs'' of CM are discouraged.
  Interventions: Procedure: Coronary angiography using conventional manual injection syringe.

INTERVENTIONS:
Device: Coronary angiography using DyeVert system — Invasive diagnostic and/or interventional cardiovascular procedures in the setting of acute coronary syndrome using DyeVert system.
  Arms: DyeVert group
Procedure: Coronary angiography using conventional manual injection syringe. — Invasive diagnostic and/or interventional cardiovascular procedures in the setting of acute coronary syndrome using conventional manual injection syringe.
  Arms: Control group

SUMMARY:
The aim of the REnal Insufficiency Following Contrast MEDIA Administration TriaL IV (REMEDIAL IV) is to test whether the use of the DyeVert system is effective in reducing CI-AKI rate in ACS patients undergoing urgent/immediate (within 2 hours) invasive diagnostic and/or interventional cardiovascular procedures. The DyeVert™ system (Osprey Medical Inc., Minnetonka, MN, USA) is a novel device designed to reduce CM volume during coronary procedures, while maintaining fluoroscopic image quality.

Patients with ACS scheduled for urgent/immediate coronary angiography/angioplasty will be enrolled and randomized into 2 groups: 1) DyeVert group (CM injection will be handled by the DyeVert TM system), and 2) Control group (CM injection will be carried out by a conventional manual injection syringe).

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication in patients suffering from acute coronary syndromes (ACS) and treated by percutaneous coronary intervention (PCI). This complication has been associated with higher early and late adverse events. It has been emphasized that the pathogenesis of AKI in the setting of ACS is multifactorial, including age, unstable hemodynamic conditions, co-morbidities (that is, diabetes mellitus and anemia) pre-existing chronic kidney disease, dehydration and administration of nephrotoxic drugs. However, the role of iodinated contrast media (CM) has been well established. Hydration represents the cornerstone in contrast-induced AKI (CI-AKI) prevention. However, at present there is no consensus on how hydration should be carried out, especially in ACS patients, and all the the recommended hydration regimens have limited applicability in the urgent/emergent settings such as ACS. Several targeted hydration regimens have been proposed, but none has been tested in ACS patients; in the present trial the investigators will adopt the left ventricular end diastolic pressure (LVEDP) -guided hydration because this approach is simple and easy to implement in the current target population. The CM volume used is an independent predictor of CI-AKI and the concept that "the lower the CM volume, the lower the CI-AKI risk" is generally accepted. The administration of a CM volume >3X glomerular filtration rate (GFR) is suggestive of increased risk of CI-AKI. To date the use of manual injections with a manifold remains the preferred technique in the majority of catheterization laboratories. In particular, manual injection is often favored for interventional procedures, which require low, variable-flow pressure injections. The AVERT trial demonstrated that CM volume is significantly lower in patients randomized to DyeVert™ in comparison to control (36.9 ± 10.9 mL versus 62.5 ± 12.7 mL, p < 0.001) and the observed reduction in CM volume used was most evident in patients undergoing PCI. Therefore, in this scenario is of outmost importance to limit the CM volume in the attempt to prevent CI-AKI. The aim of the REnal Insufficiency Following Contrast MEDIA Administration TriaL IV (REMEDIAL IV) is to test whether the use of the DyeVert system is effective in reducing CI-AKI rate in ACS patients undergoing urgent or immediate (within 2 hours) invasive diagnostic and/or interventional cardiovascular procedures.

METHODS All patients with ACS scheduled for urgent/immediate coronary angiography/angioplasty will be screened for inclusion/exclusion criteria. Diagnosis of ACS (both ST-Elevation Myocardial Infarction [STEMI] and high-risk Non-ST-Elevation Myocardial Infarction [Non-STEMI]) will be established in accordance with guidelines, including a typical chest pain history, diagnostic electrocardiographic changes, and serial increase of cardiac biomarkers. All patients with inclusion/exclusion criteria satisfied and who will agree to sign the informed consent will be enrolled into the trial. The REMEDIAL IV trial will be conducted at a pool of Italian interventional cardiology centers, according to the principles of the Declaration of Helsinki and Good Clinical Practice and has been approved by the local Ethic Committees.

All the patients included into the study will receive intravenous 0.9% sodium chloride as soon as in the catheterization laboratory; the hydration regimen will be defined according to the hemodynamic conditions, as defined below. The patients will be then randomized into 2 groups: 1) DyeVert group, and 2) Control group.

STUDY ENDPOINTS The primary endpoint of the trial is the rate of CI-AKI. CI-AKI is defined as an increase in the serum creatinine (sCr) concentration ≥ 0.3 mg/dL from the baseline value within 5 days after CM administration or the need for dialysis. Secondary end-points will include: 1) differences in the CM volume in the 2 groups; 2) an increase in the sCr concentration ≥25% within 5 days after CM exposure; 4) the severity of AKI assessed according to the Acute Kidney Injury Network criteria: Stage 1, a sCr increase ≥0.3 mg/dL or ≥1.5-1.9 times from baseline; Stage 2, a sCr increase ≥2.0-2.9 times from baseline; and Stage 3, a sCr increase ≥3.0 times from baseline or the need for dialysis; 5) changes in the serum cystatin C concentration at 24 and 48 hours after CM exposure; 6) the rate of acute renal failure requiring dialysis (defined as a decrease in renal function necessitating acute hemodialysis, ultrafiltration or peritoneal dialysis within the first 5 days post-intervention); 7) the rate of in-hospital, 6 and 12-month major adverse events (MAE), including death, renal failure requiring dialysis, acute pulmonary edema, and sustained kidney injury. Sustained kidney injury is defined as a persistent ≥25% GFR reduction compared to baseline at 6 and 12 months; and 8) the length in in-hospital stay, calculated as the sum of the number of days since admission until discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Urgent or immediate (within 2 hours) coronary procedure with iodinated contrast media administration in the setting of an acute coronary syndrome:

ST-Elevation Myocardial Infarction (according to Fourth Universal Definition of Myocardial Infarction);

High-risk Non-ST-Elevation Myocardial Infarction (according to current guidelines):

1. Refractory angina,
2. Signs or symptoms of heart faiklure or new or worsening mitral regurgitation,
3. Hemodynamic instability,
4. Recurrent angina or ischemia at rest or with low-level activities despite intensive medical therapy,
5. Sustained ventricular tachycardia or ventricular fibrillation,
6. Recurrent dynamic ST-T wave changes, particularly with intermittent ST-elevation.

Exclusion Criteria:

* Women who are pregnant.
* Recent contrast media exposure: contrast media exposure within 48 hours.
* End-stage chronic kidney disease on chronic dialysis: both haemodialysis and peritoneal dialysis.
* Multiple myeloma.
* Current enrolment in any other study when enrolment in the REMEDIAL IV would involve deviation from either protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of contrast-induced Acute Kidney Injury (CI-AKI). | 30 days
  Serum creatinine (mg(dL) is assessed at baseline (before coronary intervention) and then every day during the hospital stay. CI-AKI is defined as a change in the serum creatinine concentration ≥0.3 mg/dL from the baseline value within 5 days after contrast media administration or the need for dialysis.

SECONDARY OUTCOMES:
Differences in the contrast media volume in the 2 groups. | 30 days
  Volume of contrast media utilized (mL) is assessed in all enrolled patients at the end of the procedure
Change in the sCr concentration ≥ 25 percent within 5 days after CM exposure. | 30 days
  Serum creatinine (mg(dL) is assessed at baseline at baseline (before coronary intervention) and therefore every day during the hospidal stay
Severity of AKI assessed according to the Acute Kidney Injury Network criteria. | 30 days
  Stage 1, a sCr change ≥0.3 mg/dL or ≥1.5-1.9 times from baseline; Stage 2, a sCr change ≥2.0-2.9 times from baseline; Stage 3, a sCr change ≥3.0 times from baseline or the need for dialysis.
Changes in the serum cystatin C concentration at 24 and 48 hours after CM exposure. | 48 hours
  Serum Cystatin C (mg/dL) is assessed at baseline (before the coronary procedure) and at 24 and 48 hours after the procedure
Rate of acute renal failure requiring dialysis. | 5 days
  Change in renal function necessitating acute hemodialysis, ultrafiltration or peritoneal dialysis within the first 5 days post intervention.
Rate of in-hospital, 6 and 12 month major adverse events (MAE). | 12 months
  MAE include death, renal failure requiring dialysis, acute pulmonary edema, and sustained kidney injury (defined as a persistent ≥25% GFR change compared to baseline at 6 and 12 months
Length of in-hospital stay. | 30 days
  In-hospital stay calculated as the sum of the number of days since admission until discharge from the hospital.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Policlinico Multimedica, Milan
  - Clinica Mediterranea, Naples

REFERENCES:
- [Result] Marenzi G, Lauri G, Assanelli E, Campodonico J, De Metrio M, Marana I, Grazi M, Veglia F, Bartorelli AL. Contrast-induced nephropathy in patients undergoing primary angioplasty for acute myocardial infarction. J Am Coll Cardiol. 2004 Nov 2;44(9):1780-5. doi: 10.1016/j.jacc.2004.07.043. PMID 15519007
- [Result] Maioli M, Toso A, Leoncini M, Micheletti C, Bellandi F. Effects of hydration in contrast-induced acute kidney injury after primary angioplasty: a randomized, controlled trial. Circ Cardiovasc Interv. 2011 Oct 1;4(5):456-62. doi: 10.1161/CIRCINTERVENTIONS.111.961391. Epub 2011 Oct 4. PMID 21972403
- [Result] Giacoppo D, Madhavan MV, Baber U, Warren J, Bansilal S, Witzenbichler B, Dangas GD, Kirtane AJ, Xu K, Kornowski R, Brener SJ, Genereux P, Stone GW, Mehran R. Impact of Contrast-Induced Acute Kidney Injury After Percutaneous Coronary Intervention on Short- and Long-Term Outcomes: Pooled Analysis From the HORIZONS-AMI and ACUITY Trials. Circ Cardiovasc Interv. 2015 Aug;8(8):e002475. doi: 10.1161/CIRCINTERVENTIONS.114.002475. PMID 26198286
- [Result] Ronco C, Cicoira M, McCullough PA. Cardiorenal syndrome type 1: pathophysiological crosstalk leading to combined heart and kidney dysfunction in the setting of acutely decompensated heart failure. J Am Coll Cardiol. 2012 Sep 18;60(12):1031-42. doi: 10.1016/j.jacc.2012.01.077. Epub 2012 Jul 25. PMID 22840531
- [Result] Marenzi G, Assanelli E, Campodonico J, Lauri G, Marana I, De Metrio M, Moltrasio M, Grazi M, Rubino M, Veglia F, Fabbiocchi F, Bartorelli AL. Contrast volume during primary percutaneous coronary intervention and subsequent contrast-induced nephropathy and mortality. Ann Intern Med. 2009 Feb 3;150(3):170-7. doi: 10.7326/0003-4819-150-3-200902030-00006. PMID 19189906
- [Result] McCullough PA. Contrast-induced acute kidney injury. J Am Coll Cardiol. 2008 Apr 15;51(15):1419-28. doi: 10.1016/j.jacc.2007.12.035. PMID 18402894
- [Result] Desch S, Fuernau G, Poss J, Meyer-Saraei R, Saad M, Eitel I, Thiele H, de Waha S. Impact of a novel contrast reduction system on contrast savings in coronary angiography - The DyeVert randomised controlled trial. Int J Cardiol. 2018 Apr 15;257:50-53. doi: 10.1016/j.ijcard.2017.12.107. Epub 2018 Jan 2. PMID 29373136
- [Result] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Result] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ. 2014 AHA/ACC Guideline for the Management of Patients with Non-ST-Elevation Acute Coronary Syndromes: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Dec 23;64(24):e139-e228. doi: 10.1016/j.jacc.2014.09.017. Epub 2014 Sep 23. No abstract available. PMID 25260718
- [Result] Roffi M, Patrono C, Collet JP, Mueller C, Valgimigli M, Andreotti F, Bax JJ, Borger MA, Brotons C, Chew DP, Gencer B, Hasenfuss G, Kjeldsen K, Lancellotti P, Landmesser U, Mehilli J, Mukherjee D, Storey RF, Windecker S; ESC Scientific Document Group. 2015 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: Task Force for the Management of Acute Coronary Syndromes in Patients Presenting without Persistent ST-Segment Elevation of the European Society of Cardiology (ESC). Eur Heart J. 2016 Jan 14;37(3):267-315. doi: 10.1093/eurheartj/ehv320. Epub 2015 Aug 29. No abstract available. PMID 26320110
- [Result] Brar SS, Aharonian V, Mansukhani P, Moore N, Shen AY, Jorgensen M, Dua A, Short L, Kane K. Haemodynamic-guided fluid administration for the prevention of contrast-induced acute kidney injury: the POSEIDON randomised controlled trial. Lancet. 2014 May 24;383(9931):1814-23. doi: 10.1016/S0140-6736(14)60689-9. PMID 24856027
- [Result] Nayak KR, Mehta HS, Price MJ, Russo RJ, Stinis CT, Moses JW, Mehran R, Leon MB, Kandzari DE, Teirstein PS. A novel technique for ultra-low contrast administration during angiography or intervention. Catheter Cardiovasc Interv. 2010 Jun 1;75(7):1076-83. doi: 10.1002/ccd.22414. PMID 20146209
- [Result] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Result] Mehran R, Aymong ED, Nikolsky E, Lasic Z, Iakovou I, Fahy M, Mintz GS, Lansky AJ, Moses JW, Stone GW, Leon MB, Dangas G. A simple risk score for prediction of contrast-induced nephropathy after percutaneous coronary intervention: development and initial validation. J Am Coll Cardiol. 2004 Oct 6;44(7):1393-9. doi: 10.1016/j.jacc.2004.06.068. PMID 15464318
- [Result] Gurm HS, Seth M, Kooiman J, Share D. A novel tool for reliable and accurate prediction of renal complications in patients undergoing percutaneous coronary intervention. J Am Coll Cardiol. 2013 Jun 4;61(22):2242-8. doi: 10.1016/j.jacc.2013.03.026. PMID 23721921
- [Result] Gurm HS, Dixon SR, Smith DE, Share D, Lalonde T, Greenbaum A, Moscucci M; BMC2 (Blue Cross Blue Shield of Michigan Cardiovascular Consortium) Registry. Renal function-based contrast dosing to define safe limits of radiographic contrast media in patients undergoing percutaneous coronary interventions. J Am Coll Cardiol. 2011 Aug 23;58(9):907-14. doi: 10.1016/j.jacc.2011.05.023. PMID 21851878
- [Result] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Result] Briguori C, Quintavalle C, De Micco F, Visconti G, Di Palma V, Napolitano G, Focaccio A, Condorelli G. Persistent serum creatinine increase following contrast-induced acute kidney injury. Catheter Cardiovasc Interv. 2018 Jun;91(7):1185-1191. doi: 10.1002/ccd.27239. Epub 2017 Aug 11. PMID 28799717
- [Result] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Result] Leoncini M, Toso A, Maioli M, Tropeano F, Villani S, Bellandi F. Early high-dose rosuvastatin for contrast-induced nephropathy prevention in acute coronary syndrome: Results from the PRATO-ACS Study (Protective Effect of Rosuvastatin and Antiplatelet Therapy On contrast-induced acute kidney injury and myocardial damage in patients with Acute Coronary Syndrome). J Am Coll Cardiol. 2014 Jan 7-14;63(1):71-9. doi: 10.1016/j.jacc.2013.04.105. Epub 2013 Sep 26. PMID 24076283
- [Result] Ando G, Cortese B, Russo F, Rothenbuhler M, Frigoli E, Gargiulo G, Briguori C, Vranckx P, Leonardi S, Guiducci V, Belloni F, Ferrari F, de la Torre Hernandez JM, Curello S, Liistro F, Perkan A, De Servi S, Casu G, Dellavalle A, Fischetti D, Micari A, Loi B, Mangiacapra F, Russo N, Tarantino F, Saia F, Heg D, Windecker S, Juni P, Valgimigli M; MATRIX Investigators. Acute Kidney Injury After Radial or Femoral Access for Invasive Acute Coronary Syndrome Management: AKI-MATRIX. J Am Coll Cardiol. 2017 May 11:S0735-1097(17)36897-3. doi: 10.1016/j.jacc.2017.02.070. Online ahead of print. PMID 28528767
- [Result] Solomon R, Werner C, Mann D, D'Elia J, Silva P. Effects of saline, mannitol, and furosemide on acute decreases in renal function induced by radiocontrast agents. N Engl J Med. 1994 Nov 24;331(21):1416-20. doi: 10.1056/NEJM199411243312104. PMID 7969280
- [Result] Briguori C, Visconti G, Focaccio A, Airoldi F, Valgimigli M, Sangiorgi GM, Golia B, Ricciardelli B, Condorelli G; REMEDIAL II Investigators. Renal Insufficiency After Contrast Media Administration Trial II (REMEDIAL II): RenalGuard System in high-risk patients for contrast-induced acute kidney injury. Circulation. 2011 Sep 13;124(11):1260-9. doi: 10.1161/CIRCULATIONAHA.111.030759. Epub 2011 Aug 15. PMID 21844075
- [Result] Narula A, Mehran R, Weisz G, Dangas GD, Yu J, Genereux P, Nikolsky E, Brener SJ, Witzenbichler B, Guagliumi G, Clark AE, Fahy M, Xu K, Brodie BR, Stone GW. Contrast-induced acute kidney injury after primary percutaneous coronary intervention: results from the HORIZONS-AMI substudy. Eur Heart J. 2014 Jun 14;35(23):1533-40. doi: 10.1093/eurheartj/ehu063. Epub 2014 Mar 6. PMID 24603308
- [Result] Naidu SS, Aronow HD, Box LC, Duffy PL, Kolansky DM, Kupfer JM, Latif F, Mulukutla SR, Rao SV, Swaminathan RV, Blankenship JC. SCAI expert consensus statement: 2016 best practices in the cardiac catheterization laboratory: (Endorsed by the cardiological society of india, and sociedad Latino Americana de Cardiologia intervencionista; Affirmation of value by the Canadian Association of interventional cardiology-Association canadienne de cardiologie d'intervention). Catheter Cardiovasc Interv. 2016 Sep;88(3):407-23. doi: 10.1002/ccd.26551. Epub 2016 May 2. No abstract available. PMID 27137680
- [Result] Hwang JR, D'Alfonso S, Kostuk WJ, Diamantouros P, Teefy P, Jablonsky G, Lavi S. Contrast volume use in manual vs automated contrast injection systems for diagnostic coronary angiography and percutaneous coronary interventions. Can J Cardiol. 2013 Mar;29(3):372-6. doi: 10.1016/j.cjca.2012.11.023. Epub 2013 Jan 24. PMID 23352426
- [Result] Mehran R, Faggioni M, Chandrasekhar J, Angiolillo DJ, Bertolet B, Jobe RL, Al-Joundi B, Brar S, Dangas G, Batchelor W, Prasad A, Gurm HS, Tumlin J, Stone GW. Effect of a Contrast Modulation System on Contrast Media Use and the Rate of Acute Kidney Injury After Coronary Angiography. JACC Cardiovasc Interv. 2018 Aug 27;11(16):1601-1610. doi: 10.1016/j.jcin.2018.04.007. PMID 30139467
- [Result] Sadick V, Reed W, Collins L, Sadick N, Heard R, Robinson J. Impact of biplane versus single-plane imaging on radiation dose, contrast load and procedural time in coronary angioplasty. Br J Radiol. 2010 May;83(989):379-94. doi: 10.1259/bjr/21696839. Epub 2009 Dec 17. PMID 20019175
- [Result] Mariani J Jr, Guedes C, Soares P, Zalc S, Campos CM, Lopes AC, Spadaro AG, Perin MA, Filho AE, Takimura CK, Ribeiro E, Kalil-Filho R, Edelman ER, Serruys PW, Lemos PA. Intravascular ultrasound guidance to minimize the use of iodine contrast in percutaneous coronary intervention: the MOZART (Minimizing cOntrast utiliZation With IVUS Guidance in coRonary angioplasTy) randomized controlled trial. JACC Cardiovasc Interv. 2014 Nov;7(11):1287-93. doi: 10.1016/j.jcin.2014.05.024. Epub 2014 Oct 15. PMID 25326742
- [Result] Gurm HS, Seth M, Mehran R, Cannon L, Grines CL, LaLonde T, Briguori C; Blue Cross Blue Shield of Michigan Cardiovascular Consortium (BMC2). Impact of Contrast Dose Reduction on Incidence of Acute Kidney Injury (AKI) Among Patients Undergoing PCI: A Modeling Study. J Invasive Cardiol. 2016 Apr;28(4):142-6. Epub 2016 Jan 15. PMID 26773238
- [Result] Freeman RV, O'Donnell M, Share D, Meengs WL, Kline-Rogers E, Clark VL, DeFranco AC, Eagle KA, McGinnity JG, Patel K, Maxwell-Eward A, Bondie D, Moscucci M; Blue Cross-Blue Shield of Michigan Cardiovascular Consortium (BMC2). Nephropathy requiring dialysis after percutaneous coronary intervention and the critical role of an adjusted contrast dose. Am J Cardiol. 2002 Nov 15;90(10):1068-73. doi: 10.1016/s0002-9149(02)02771-6. PMID 12423705
- [Result] Qian G, Fu Z, Guo J, Cao F, Chen Y. Prevention of Contrast-Induced Nephropathy by Central Venous Pressure-Guided Fluid Administration in Chronic Kidney Disease and Congestive Heart Failure Patients. JACC Cardiovasc Interv. 2016 Jan 11;9(1):89-96. doi: 10.1016/j.jcin.2015.09.026. Epub 2015 Dec 9. PMID 26685074
- [Derived] Briguori C, Quintavalle C, Mariano E, D'Agostino A, Scarpelli M, Focaccio A, Zoccai GB, Evola S, Esposito G, Sangiorgi GM, Condorelli G. Kidney Injury After Minimal Radiographic Contrast Administration in Patients With Acute Coronary Syndromes. J Am Coll Cardiol. 2024 Mar 19;83(11):1059-1069. doi: 10.1016/j.jacc.2024.01.016. PMID 38479953